CLINICAL TRIAL: NCT03222752
Title: A 6 Week, Randomized, Double-blind, Placebo Controlled Trial of the Efficacy and Tolerability of Cranial Electrotherapy Stimulation for the Treatment of Major Depressive Disorder, With a 6 Week Open Label Extension Phase.
Brief Title: Efficacy of Cranial Electrotherapy Stimulation (CES) for the Treatment of Major Depressive Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant recruitment insufficient to complete study
Sponsor: Electromedical Products International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MDD1
Record Dates: First submitted 2017-06-19; First posted 2017-07-19 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Major Depressive Disorder
Keywords: Alpha-Stim; Cranial Electrotherapy Stimulation; CES
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: A single site, 6 week, randomized, double-blind, placebo controlled evaluation of efficacy and tolerability of cranial electrotherapy stimulation (CES) for the treatment of adults from 18-65 years of age with treatment resistant Major Depressive Disorder (MDD) with a 6 week open label extension phase.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatment device will deliver subsensory treatment while the sham device will deliver no treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Group (Active Comparator): Group receives active treatment for 6 weeks. The intervention used will be cranial electrotherapy stimulation from and Alpha-Stim AID.
  Interventions: Device: Cranial Electrotherapy Stimulation
- Sham Treatment Group (Sham Comparator): Groups receives treatment using sham cranial electrotherapy stimulation devices for 6 weeks. No actual treatment will be received. This group will not receive any treatment interventions. The same outcome measures will be used as the treatment group.
  Interventions: Device: Sham Cranial Electrotherapy Stimulation

INTERVENTIONS:
Device: Cranial Electrotherapy Stimulation — Alpha-Stim® AID microcurrent and cranial electrotherapy stimulator will be used. Daily one hour cranial electrotherapy stimulation (CES) treatment using ear clip electrodes with current set at fixed level of 100 uA (a subsensory current level), 0.5 Hertz will be used for active CES treatment group for 6 weeks. For the sham group the Alpha-Stim® AID ear clips will not emit electricity.
  Other Names: Alpha-Stim
  Arms: Treatment Group
Device: Sham Cranial Electrotherapy Stimulation — The sham treatment will be using a sham Alpha-Stim AID which will look and sound exactly like the active treatment but will deliver no current.
  Other Names: Sham Alpha-Stim
  Arms: Sham Treatment Group

SUMMARY:
Efficacy of Cranial Electrotherapy Stimulation (CES) for the treatment of Major Depressive Disorder

DETAILED DESCRIPTION:
A 6 week, randomized, double-blind, placebo controlled trial of the efficacy and tolerability of Cranial Electrotherapy Stimulation for the treatment of Major Depressive Disorder, with a 6 week open label extension phase.

ELIGIBILITY:
Inclusion Criteria:

Patients must be able to provide informed consent and sign the informed consent form prior to the conduct of any study specific procedures. To be eligible to participate in the study, patients must meet the following criteria:

1. Subject is a male or female outpatient age 22 to 65 years, inclusive.
2. Subject meets DSM-5 criteria for MDD as determined by MINI screening interview.
3. The subject has a score of > 4 on CGI-S on visit 1 and 2.
4. Sexually active female patients of childbearing potential must be practicing at least one or more the following methods of contraception during the study: intrauterine device (IUD), barrier method in combination with a spermicide, oral/hormonal contraception or abstinence. Female patients of childbearing potential must have a negative pregnancy test prior to receiving study treatment.
5. Subject is in good medical health or with chronic medical conditions which are currently stable.
6. No current abuse of alcohol or other substance.
7. Capable of doing active or sham CES treatments and completing all study requirements independently.
8. The subject has a score of ≥ 17 on the HAM-D. If a subject is being treated with Serotonin Selective Reuptake Inhibitor (SSRIs) medications which include: Fluoxetine (Prozac), Paroxetine (Paxil), Sertraline (Zoloft), Luvox (Fluvoxamine), Citalopram (Celexa) and Escitalopram (Lexapro), as well as serotonin and norepinephrine reuptake inhibitors (SNRI) such as Venlafaxine (Effexor IR and XR), Desvenlafaxine (Pristiq) and Duloxetine (Cymbalta) they may remain on one of the SSRI or SNRI medications provided that he or she has been on a stable dose for at least 4 weeks prior to entering this study; this dose is to remain stable throughout the remainder of this study (any need to change the dose during the study will be evaluated and will result in termination).

Exclusion Criteria:

Patients will be not be considered for inclusion into the study if they meet any of the conditions below:

1. Subject meets DSM-5 criteria for another axis 1 disorder (other than MDD) as the primary diagnosis (i.e., schizophrenia, mood disorder, psychosis, anorexia nervosa) as determined by the MINI. Conduct and antisocial personality disorders will not be allowed to participate. Patients with comorbid diagnoses of learning disorders, attention deficit disorder (with or without hyperactivity), communication disorders, separation anxiety disorder, dysthymic disorder or anxiety disorders will be allowed to participate in the study as long as these conditions are not the primary focus of any treatment and they comply with concomitant medication limitations listed in the appendix. Those with substance use disorders will not be allowed to participate.
2. Subject is clinically judged by the investigator to be at risk for suicide or is acutely suicidal as objectively measured by the C-SSRS.
3. Subject has attempted suicide one or more times within the past 12 months
4. Subject has a Hamilton Depression Rating Scale17 (HAM-D17) score above 38 which suggests a moderate to severe clinical level of depressive symptoms
5. Subject has a psychiatric condition that would require inpatient, or partial psychiatric hospitalization.
6. There is an imminent risk of injuring self or others or causing damage to property as judged by the investigator.
7. Subject has a significant history of medical disease (i.e., cardiovascular, hepatic (e.g., cirrhosis, hepatitis B or C) renal, gynecological, musculoskeletal, neurological, gastrointestinal, metabolic, hematological, endocrine, cancer with a metastatic potential, progressive neurological disorders or seizure disorder) which could impair reliable participation in the trial or necessitate the use of medication not allowed by this protocol unless all of the following are true (consultation with study physician is encouraged before patient enrollment):

   1. The condition has been stable for over one year (3 years for malignancy other than excised basal cell carcinoma, for which one year stability is required).
   2. The condition has been judged by the Investigator not to interfere with the patient's participation in the study.
   3. The condition is fully documented in the patient's study records.
8. Hypo- or hyperthyroidism, unless stabilized on appropriate pharmacotherapy with no change in dosage for at least three months before visit 1 (Screening).
9. Subject is pregnant, planning to become pregnant, or nursing. If a subject becomes pregnant, she will be discontinued immediately and followed appropriately.
10. For females who are sexually active:

    Not practicing a reliable method of contraception that will continue for the duration of the study and within 30 days following the end of study participation.

    Reliable contraception is defined as:
    1. surgical sterilization
    2. oral contraceptives (consisting of an estrogen-progestin combination or progestin alone
    3. transdermally derived contraceptives (e.g., Ortho - Evra), depot injections (e.g., Depo-Provera)
    4. vagina contraceptive ring (e.g., Nucaring), contraceptive implants (e.g., Implanon, Norplant 2/Jadelle)
    5. an intrauterine device
    6. diaphragm plus condom (the only acceptable double barrier method)
    7. other forms of contraceptives (pharmacological and/or non-pharmacological) are not accepted
11. Subject has had concomitant therapy with another investigational drug, or participation in an investigational drug study within one month prior to entering this study.
12. Subject who has initiated or terminated psychotherapy or behavior therapy within one month before visit 1 (screening), or who plans to initiate or change such therapy during the course of the study.
13. Subject has history of poor compliance or in the Investigator's opinion any subject whose treatment as an outpatient would be clinically contraindicated.
14. Subject has had previous trial of cranial electrotherapy stimulation (CES).
15. Subject requiring prohibited concomitant medication or herbal supplements that could not be discontinued or switched to an allowable alternative medication and stabilized for at least two weeks preceding (visit 2).
16. Subject taking any psychoactive drug or herbal remedy within 5 half-lives before baseline (visit 2), (St. John's wort, ginkgo biloba, kava kava, valerian root, DHEA, tyrosine, tryptophan and 5-HTP, antidepressants, anxiolytics, monoamine oxidase inhibitors, antipsychotics, or anticonvulsants/mood stabilizers, carbamazepine, or others). Patients who have ever been treated with the depot antipsychotic must also be excluded.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale | 6 weeks
  The Hamilton Rating Scale for Depression (HRSD), also called the Hamilton Depression Rating Scale (HDRS), abbreviated HAM-D, is a multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity of Illness | 6 weeks
  The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
Clinical Global Impression - Global Improvement | 6 weeks
  The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Barclay, PhD, Principal Investigator — Liberty University
Locations (1):
- Advanced Psychotherapeutics, Forest, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
PI will maintain all patient data during the trial. Data will be de identified and encrypted before sending to the designated statistician.